CLINICAL TRIAL: NCT03202511
Title: Assessment of a New "Boosting" Strategy for HIV Pre-exposure Prophylaxis in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Zeruesenay Desta, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1705315090
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Pre-Exposure Prophylaxis
MeSH Terms: interventions — Probenecid; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated to enter the study in either the control or treatment arm using a blocked design to ensure equal numbers of subjects in each sequence group (n=8, control to treatment; n=8, treatment to control). Following a washout period of at least 6 weeks, each individual will crossover to the next study phase. The randomization table will be constructed prior to subject enrollment by the Principal Investigator using the Statistical Analysis Software (SAS®) randomization procedure. In the event that an individual is withdrawn from the study, an alternate participant will replace that individual using an identical study sequence to maintain the block design. A total of 16 subjects will be initially enrolled in an effort to ensure that at least 14 subjects complete the entire study. If needed, additional subjects will be screened and enrolled until the target enrollment of n=14 subjects have completed the entire study.
Masking Description: This will be an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): The control phase will consist of subjects taking 600/400 mg oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) on day 1 (2 tablets) followed by 300/200 mg (1 tablet) doses on days 2 and 3.
  Interventions: Drug: Tenofovir disoproxil fumarate/Emtricitabine
- Treatment (Experimental): The treatment phase will consist of subjects taking 600/400 mg oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) (2 tablets) along with a 2 gram oral probenecid (PRO) dose (4 tablets, 500 mg each) on day 1.
  Interventions: Drug: Probenecid Oral Tablet; Drug: Tenofovir disoproxil fumarate/Emtricitabine

INTERVENTIONS:
Drug: Probenecid Oral Tablet — Included in arm/group descriptions.
  Arms: Treatment
Drug: Tenofovir disoproxil fumarate/Emtricitabine — Included in arm/group descriptions.
  Other Names: TDF/FTC, Truvada

SUMMARY:
The study will be a randomized, open-label, cross-over clinical pharmacokinetic trial to investigate a strategy for probenecid "boosting" in the setting of tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC) for HIV pre-exposure prophylaxis (PrEP). The study will be conducted at the Indiana University Clinical Research Center. All samples will be processed and the amount of tenofovir/FTC in plasma, blood, and urine, and tenofovir diphosphate and emtricitabine in peripheral blood mononuclear cells will be determined using validated analytical methods developed by the investigators at the University of Colorado. Probenecid plasma and urine concentrations will also be measured using an in-house assay. Following completion of the study, the secondary aim will be accomplished via analysis of selected samples collected at baseline and following treatment. Those selected samples will be assessed for urinary markers of proximal tubulopathy (urine total protein, albumin, creatinine, phosphorus, retinol binding protein, and beta-2-microglobulin) and serum alkaline phosphatase, osteocalcin, procollagen type 1 N propeptide, cystatin C, and creatinine to determine if the probenecid boosting strategy does indeed lead to less potential renal and bone toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 55 years old healthy (as decided from a pre-enrollment screening session described above) male participants within 32% of their ideal body weight.
2. Individuals who agree to refrain from taking any prescriptions medications, over-the-counter medications (including salicylates/aspirin), hormonal agents, and herbal, dietary, and alternative supplements that may interact with the metabolism of those study drugs at least 2 weeks prior to the start of the study and until study completion.
3. Nonsmoker or individuals willing to refrain from smoking or use of tobacco or marijuana for at least one month prior to and until the completion of the study (the entire study lasts for approximately 49 days).

Exclusion Criteria:

* 1. Are underweight (weigh less than 52 kg or 114 lb) or overweight [body mass index (BMI) greater than 32].

  2. Females will be excluded to reduce study variability for this first proof of concept study.

  3. Have insufficient renal function (estimated Creatinine Clearance ≤ 90 mL/min).

  4. Have history of current alcohol or drug abuse (more than 4 alcoholic drinks per day on a regular basis).

  5. Have history of intolerance, allergic reactions (e.g. rash) or other forms of hypersensitivities to any of the study medications (tenofovir disoproxil fumarate/ emtricitabine, probenecid).

  6. Have taken TDF or FTC as part of pre-exposure prophylaxis within the past 6 weeks.

  7. Any current major illness or chronic illness such as (but not limited to) kidney disease, hepatic disease, diabetes mellitus, gout, hypertension, coronary artery disease, chronic obstructive pulmonary disease, cancer, chronic active hepatitis B virus (HBV) infection, or HIV.

  8. History of anemia or any other significant hematologic disorder. 9. Have history or current gastrointestinal disorders such as persistent diarrhea or malabsorption that would interfere with the absorption of orally administered drugs.

  10. Have a serious infection within the last week before study enrollment. 11. Have donated blood within the past two months. 12. Have blood results that do not fall in a healthy range (e.g., blood hemoglobin less than 12.0 mg/dl).

  13. Are taking on regular basis substances that may interfere with the metabolism (breakdown) of study medications by the body, including prescription medications, over-the-counter, herbal or dietary supplements, alternative medications, or hormonal agents (i.e. oral contraceptives, intra-uterine device with hormones).

  14. Have a life style that places subjects at a higher risk for contracting HIV during the study period (e.g. active illicit drug use, excessive alcohol drinking, sexually transmitted infection (including gonorrhea, chlamydia, syphilis, herpes, human papilloma virus) within the past one year, or having more than one sexual partner in the past 6 months).

  15. Positive HIV antibody test. 16. Positive HBV surface antigen test. 17. Have participation in a research study or use of an investigational drug in the last one month.

  18. Are employed or are student under supervision of any of the investigators of this study.

  19. Cannot state a good understanding of this study including risks and requirements; are unable to follow the rules of this study.

  20. Cannot commit the time requested for this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male healthy volunteers will be enrolled.
Enrollment: 15 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon T Gufford, PharmD, PhD, Principal Investigator — Indiana Unversity School of Medicine
Locations (1):
- Indiana University Clinical Research Center at University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment TDF/FTC+PRO Dose First, Then Control TDF/FTC: Participants received the treatment phase of 600/400 mg oral TDF/FTC along with a 2 gram oral PRO on day 1, 2-week washout, then the control phase of 600/400 mg oral TDF/FTC on day 1 followed by 300/200 mg oral TDF/FTC on days 2 and 3.
- Control TDF/FTC First, Then Treatment TDF/FTC+PRO Dose: Participants received the control phase of 600/400 mg oral TDF/FTC on day 1 followed by 300/200 mg oral TDF/FTC on days 2 and 3, 2-week washout, then the treatment phase of 600/400 mg oral TDF/FTC along with a 2 gram oral PRO on day 1.
Period: Overall Study
Arm/Group | Treatment TDF/FTC+PRO Dose First, Then Control TDF/FTC | Control TDF/FTC First, Then Treatment TDF/FTC+PRO Dose
Started | 8 | 7
Completed | 7 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants received control and/or treatment phase
  The control phase will consist of subjects taking 600/400 mg oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) on day 1 (2 tablets) followed by 300/200 mg (1 tablet) doses on days 2 and 3.
  The treatment phase will consist of subjects taking 600/400 mg oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) (2 tablets) along with a 2 gram oral probenecid (PRO) dose (4 tablets, 500 mg each) on day 1.
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 26 [18 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Plasma TFV AUC0-INF GMR
Description: The geometric mean ratio (GMR) of the plasma TFV area under the curve (AUC) comparing the test phase (T) to control phase (C) was assessed. PK samples were collected from 0 to 72 hours post-dose.
Time Frame: The first 72 hours of each phase.
Population: Primary result was performed for geometric mean ratio of treatment phase to control phase.
Measure: Least Squares Mean (90% Confidence Interval); unit: ng*h/mL
Groups:
- Treatment Phase: The treatment phase will consist of subjects taking 600/400 mg oral TDF/FTC along with a 2 gram oral PRO dose on day 1.
- Control Phase: The control phase will consist of subjects taking 600/400 mg oral TDF/FTC on day 1 followed by 300/200 mg TDF/FTC on days 2 and 3.
Arm/Group | Treatment Phase | Control Phase
Number analyzed (Participants) | 14 | 14
ng*h/mL | 8.75 [8.66 to 8.84] | 8.27 [8.18 to 8.36]
Statistical Analysis 1: Comparison: Treatment Phase vs Control Phase; Test type: Equivalence — 0.8 to 1.25 equivalence margin was used; Geometric Mean Ratio = 1.61, 90% CI 2-sided [1.47 to 1.77]

2. Primary Outcome: PBMC TFV-DP AUC GMR
Description: The geometric mean ratio (GMR) of the PBMC TFV-DP area under the curve (AUC) comparing the test phase (T) to control phase (C) was assessed. PK samples were collected from 0 to 72 hours post-dose.
Time Frame: The first 72 hours of each phase.
Measure: Least Squares Mean (90% Confidence Interval); unit: fmol*h/10^6cells
Arm/Group | Treatment Phase | Control Phase
Number analyzed (Participants) | 14 | 14
fmol*h/10^6cells | 7.12 [6.96 to 7.29] | 7.38 [7.22 to 7.54]
Statistical Analysis 1: Comparison: Treatment Phase vs Control Phase; Test type: Equivalence — 80 to 125% equivalence margin was used; Geometric Mean Ratio = 77.4, 90% CI 2-sided [61.4 to 97.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 1 year during study conduction.
Description: All adverse events reported from participant were included and graded for severity by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). Adverse events were reviewed per patient by treatment and was not separated individually.
Groups:
- Control Phase: The control phase consisted of subjects taking 600/400 mg oral TDF/FTC on day 1 followed by 300/200 mg TDF/FTC on days 2 and 3.
- Treatment Phase: The treatment phase consisted of subjects taking 600/400 mg oral TDF/FTC followed by 2 gram oral PRO on day 1.
Arm/Group | Control Phase | Treatment Phase
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 2/14 | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Phase (N=14) | Treatment Phase (N=15)
Nausea, vomiting, or GERD (Gastrointestinal disorders) | 2 (2) | 8 (8)
Headache or loss of appetite (Nervous system disorders) | 2 (2) | 5 (5)
Nose bleed (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03202511/Prot_SAP_000.pdf